CLINICAL TRIAL: NCT04735081
Title: SPONDYL'UP : Prolonged Bed Rest Versus Early Raising in Vertebral Osteomyelitis - A Restrospective, Monocenter, Before/After Practice Change Study
Brief Title: Prolonged Bed Rest Versus Early Raising in Vertebral Osteomyelitis
Acronym: SPONDYL'UP
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, Medical doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI189
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Infectious; Spondylitis
Keywords: Infectious vertebral osteomyelitis; Spondylodiscitis; Bed Rest; Early Raising; Verticalization; Immobilization
MeSH Terms: conditions — Communicable Diseases; Spondylitis; Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- First group before practice change: Infectious spondylodiscitis when prolonged immoblization in bed was recommanded in our hospital
- Second group after practice change: Infectious spondylodiscitis when early verticalization was recommanded in our hospital

SUMMARY:
Infectious vertebral osteomyelitis are infectious diseases of the vertebral bone, intervertebral disc and/ or adjacent tissue. Most of cases are due to hematogenous dissemination of pathogen but direct inoculation is an aetiology after surgery. Majority of cases concern adults after 50 years and the annual incidence ranging between 0.5 and 2.4 cases per 100 000 habitants in Europe but seems to increase during last 20 years.

The infectious spondylodiscitis is an important source of morbidity and mortality. The treatment is based on pathogen adapted antimicrobial therapy, which may be associated with bedrest. Surgical act is necessary when neurological complication occurs or when vertebral column instability is too important. The immobilization in bed is use to limit pain and neurological complications. However, the immobilization is based on few literature data and causes important complications especially in elderly.

The of immobilization in Nancy universitity hospital changed in 2019 after institutional recommendations based on expert opinion which recommend an early verticalization of uncomplicated spondylodiscitis. The investigators aimed to evaluate the consequences of this practice change on the hospitalization duration and complication rates due to spondylodiscitis and immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Infectious spondylodiscitis proven by radiological exam
* Infectious spondylodiscitis with microbiological documentation

Exclusion Criteria:

* Patient included in COROSIVE study
* Vertebral prosthetic device infection
* Infectious spondylodiscitis relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite infectious spondylodiscitis hospitalised between 2016 and 2022 in Nancy University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | when the patient is discharged from hospital (up to 52 weeks)
  Duration between first and last day of hospitalisation in days

SECONDARY OUTCOMES:
Rate of neurological complications | During hospitalisation (up to 52 weeks)
  Measurement of the rate spondylodiscitis-related neurological complications in each group during hospitalisation

OTHER OUTCOMES:
Rate of immobilization complications | During hospitalisation (up to 52 weeks)
  Measurement of the rate of bedrest complications in each group during hospitalisation
Mortality | During hospitalisation (up to 52 weeks)
  Patient death